CLINICAL TRIAL: NCT01319422
Title: Clinical and Pharmacodynamic Comparison of Continuous Versus Intermittent Dosing Regimens for Pomalidomide in Relapsed/Refractory Multiple Myeloma
Brief Title: Continuous Versus Intermittent Dosing Regimens for Pomalidomide in Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC 1011007607
Record Dates: First submitted 2011-03-14; First posted 2011-03-21 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Myeloma
Keywords: myeloma; multiple myeloma; pomalidomide; immunomodulatory
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pomalidomide 2 mg/d on 28 days/28 day cycle (Experimental)
  Interventions: Drug: Pomalidomide
- Pomalidomide 4 mg/d on 21 days/28 day cycle (Experimental)
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — Comparison of different dosages and schedules of drug
  Other Names: CC-4047

SUMMARY:
Lenalidomide has clinical activity in myeloma. The closely related compound, Pomalidomide, may have clinical activity in patients who have previously been treated with lenalidomide and who no longer respond to it. The mechanism of anti-tumor effects of these drugs has been attributed to several effects including anti-angiogenesis, immune activation, and anti-proliferative effects. Recent studies have suggested that these agents can mediate surprisingly rapid biologic effects on human monocytes and T cells. Our hypothesis is that the proximate effects of these drugs will be sensitive and quantitative surrogates of subsequent effects including activation of tumor antigen specific T cells as well as innate immune cells. Understanding the correlation between the pharmacodynamics of these effects with downstream activation using quantitative assays will facilitate the rational development of pomalidomide as immune-modulatory drug in diverse settings as well as its optimal development in myeloma therapy.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a common hematologic malignancy characterized by clonal expansion of transformed plasma cells (PCs) in the bone marrow1. Over the past decade, the introduction of immunomodulatory agents (such as thalidomide and lenalidomide) and proteasome inhibitors (such as bortezomib) as effective therapies has altered the therapeutic landscape for multiple myeloma (MM). Following the approval and establishment of thalidomide-containing regimens, such as melphalan, prednisone and thalidomide (MPT) and Thal/Dex, as the standard first-line therapy for newly diagnosed MM (NDMM), lenalidomide in combination with dexamethasone (RD) was approved for the treatment of patients with previously treated multiple myeloma 1 (MM1). However, even with these newly approved agents, MM remains an incurable disease and most patients will eventually relapse and progress after multiple lines of different therapeutic regimens including both lenalidomide as well as bortezomib. Thus there remains a continued need to identify newer agents to maintain long term disease control in these patients.

Thalidomide and its immune-modulatory analogue lenalidomide have clinical activity in myeloma. Pomalidomide, a thalidomide analogue, is an immunomodulatory agent that displays similar anti-angiogenic activity, but far greater anti-proliferative and immunomodulatory activity, compared to the parent drug. Pomalidomide and lenalidomide have been shown to possess very similar pharmacological properties in vitro, including anti-angiogenic, immunomodulatory and anti-proliferative properties. However a unifying molecular mechanism for these diverse effects has been elusive. Pomalidomide and lenalidomide have significantly greater capacity for enhanced costimulation, leading to enhanced activation of innate and adaptive immune cells compared to Thalidomide. Recent studies have yielded the surprising finding that these agents can mediate rapid biologic effects on human monocytes and T cells in culture leading to activation of ras homolog gene family, member A (RhoA) GTPases, and enhanced actin polymerization. Changes in actin cytoskeleton may also contribute to the capacity to these drugs to enhance the formation of immune synapses, Pomalidomide has also been shown to stimulate antibody-dependent cytotoxic T-cell activity (ADCC) in preclinical models.

At tolerated doses (MTD = 2 mg per day (QD) and 5 mg every other day (QOD), pomalidomide has been shown to be active in subjects with relapsed or refractory multiple myeloma (study CC-4047-00-001). In 45 subjects who received doses of pomalidomide ranging, by cohort, up to 10 mg daily, the most commonly occurring dose-limiting toxicity (DLT) was reversible neutropenia. As with other immunomodulatory drugs (IMiDs) administered to subjects receiving concomitant systemic steroids, deep vein thrombosis (DVT) was seen (in 1 subject each in this study and in its subsequent named patient supply rollover program).

Recently, preliminary efficacy and safety data from an ongoing phase II study, led by Martha Lacy at Mayo Clinic, were published. Sixty patients with relapsed or refractory multiple myeloma were enrolled. Pomalidomide (CC-4047) was given orally at a dose of 2 mg daily on days 1-28 of a 28-day cycle and dexamethasone was given orally at a dose of 40 mg daily on days 1, 8, 15, 22 of each cycle. Patient also received aspirin 325 mg once daily for thromboprophylaxis. The study endpoints were the response rate in patients taking pomalidomide plus dexamethasone including patients with lenalidomide resistant refractory multiple myeloma, and safety of pomalidomide plus dexamethasone. Responses were recorded using the criteria of the International Myeloma Working Group. Thirty eight patients achieved objective response (63%) including complete response (CR) in 3 patients (5%), very good partial response (VGPR) in 17 patients (28%), and partial response (PR) in 18 patients (30%). The CR + VGPR rate was 33%. Grade 3 or 4 hematologic toxicity occurred in 23 patients (38%) and consisted of anemia in three patients (5%), thrombocytopenia in two patients (3%) and neutropenia in 21 (35%). Among those that developed grade 3/4 neutropenia, all first experienced the neutropenia in cycle 1-3; no new patients experienced grade 3/4 neutropenia in cycle 4 or later. The most common non-hematological grade 3/4 toxicities were fatigue (17%) and pneumonia (8%). Other grade 3/4 non-hematological toxicities that occurred in less than 5% included diarrhea, constipation, hyperglycemia, and neuropathy. One patient (1.6%) had a thromboembolic event of deep vein thrombosis.

Another dosing regimen for Pomalidomide involved 21/28 day dosing, as in the current dosing regimen for Lenalidomide. In this trial the recommended dose for phase II testing was determined to be 4 mg, 21/28 d. Clinical response (greater than or equal to a partial response (PR)) was observed in 7/25 (28%) patients. While both regimens seem to be clinically active, it is unclear at present as to which regimen leads to greater immune activation or clinical activity.

In addition to MM, pre-clinical data and the prior experience with thalidomide and lenalidomide in the treatment of patients with myelofibrosis with myeloid metaplasia (MMM) provided the rationale for the use of pomalidomide in patients with MMM. This is further supported by the results of a Celgene sponsored trial (MMM-001) which indicated that pomalidomide therapy at 0.5 mg or 2 mg/day +/- an abbreviated course of prednisone is well tolerated in patients with myelofibrosis and active in the treatment of anemia.

However, these studies did not monitor proximate pharmacodynamic events (such as might occur within hours of drug exposure), and link these to downstream effects, including clinical activity and toxicity. Our hypothesis is that the proximate effects of these drugs (including drug induced changes in F-actin) and early phosphorylation events will be sensitive and quantitative surrogates of subsequent effects including activation of tumor antigen specific T cells as well as innate immune cells. Understanding the correlation between pharmacodynamics of these effects with downstream activation using quantitative assays will facilitate rational development of these agents as immunomodulatory drugs in diverse settings and may also allow optimization of drug delivery to both reduce potential toxicity, and enhance efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age ≥18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Relapsed / Refractory Multiple Myeloma following at least two prior standard therapies including lenalidomide. Induction therapy followed by autologous stem cell transplantation (ASCT) is considered one regimen.
* Patients must be refractory to prior lenalidomide therapy. For the purpose of this protocol, refractory will be defined as history of progression on a regimen containing full or maximally tolerated dose of lenalidomide administered for a minimum of at least one complete cycle of therapy.
* All patients must have measurable disease defined as one or more of the following criteria:

  * Serum monoclonal protein greater than 10 g/L, serum immunoglobulin free light chain (FLC) more than 10 mg/dL and an abnormal FLC ratio, urine light-chain excretion > 200 mg/24 h, measurable soft tissue plasmacytoma that has not been irradiated, or greater than 30% plasma cells in bone marrow.
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 2 weeks prior to treatment in this study.
* Eastern Cooperative Oncology Group (ECOG ) performance status of ≤ 2 at study entry (see Appendix D).
* Laboratory test results within these ranges:

  * Absolute neutrophil count ≥ 1.0 x 1000/microliter (uL)
  * Platelet count ≥ 75 x 1000/uL
  * Serum creatinine ≤ 2.5 mg/dL
  * Total bilirubin ≤ 2 mg/dL
  * aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) ≤ 5 x upper limit of normal (ULN)
* Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 milli-international unit (mIU)/mL within 10 - 14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix A and B: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, AND also Education and Counseling Guidance Document.
* Able to take aspirin (ASA) (81 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking pomalidomide).
* Women of child-bearing potential who are unwilling to use a dual method of contraception; and men who are unwilling to use a condom.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide or lenalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, pomalidomide or similar drugs.
* Any prior use of pomalidomide.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or active infectious hepatitis, B or C.
* Grade 3 or 4 peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Dhodapkar, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Sehgal K, Das R, Zhang L, Verma R, Deng Y, Kocoglu M, Vasquez J, Koduru S, Ren Y, Wang M, Couto S, Breider M, Hansel D, Seropian S, Cooper D, Thakurta A, Yao X, Dhodapkar KM, Dhodapkar MV. Clinical and pharmacodynamic analysis of pomalidomide dosing strategies in myeloma: impact of immune activation and cereblon targets. Blood. 2015 Jun 25;125(26):4042-51. doi: 10.1182/blood-2014-11-611426. Epub 2015 Apr 13. PMID 25869284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at an academic medical center.
Pre-assignment Details: Four screened subjects did not meet eligibility criteria. Forty subjects were enrolled, but one withdrew after randomization without receiving treatment, and is listed as a "non-completer". Thus, data are presented for 39 participants.
Period: Overall Study
Arm/Group | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Median (Full Range); unit: years] | 63 [44 to 87] | 61 [47 to 80] | 61 [44 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 10 | 12 | 22
Immunoglobulin Heavy chain (IgH) type [Number; unit: participants]
  Immunoglobulin G (IgG) | 8 | 12 | 20
  Immunoglobulin A (IgA) | 4 | 1 | 5
  Light chain only | 7 | 7 | 14
Immunoglobulin Light chain (IgL) type [Number; unit: participants]
  kappa | 13 | 15 | 28
  lambda | 6 | 5 | 11
serum beta 2 microglobulin [Mean (Full Range); unit: mg/L] | 3.0 [1.55 to 5.12] | 3.4 [2.09 to 8.36] | 3.2 [1.55 to 8.36]
serum albumin [Mean (Full Range); unit: g/dL] | 3.9 [3.2 to 5.0] | 3.9 [3.2 to 4.8] | 3.9 [3.2 to 5.0]
lines of prior therapy [Median (Full Range); unit: lines] | 4 [2 to 7] | 4 [2 to 9] | 4 [2 to 9]
Deletion of chromosome 17p [Number; unit: participants]
  yes | 4 | 3 | 7
  no | 10 | 9 | 19
  missing | 5 | 8 | 13
Chromosome 1q abnormalities [Number; unit: participants]
  yes | 10 | 8 | 18
  no | 9 | 12 | 21
Deletion chromosome 13 [Number; unit: participants] — Monosomy 13 on molecular cytogenics or deletion of 13q on fluorescence in situ hybridization (FISH) cytogenics
  participants
    yes | 5 | 8 | 13
    no | 14 | 12 | 26
Lenalidomide (Len) as most recent therapy [Number; unit: participants]
  yes | 6 | 9 | 15
  no | 13 | 11 | 24
Resistance to prior therapy-Len refractory [Number; unit: participants]
  yes | 19 | 20 | 39
  no | 0 | 0 | 0
Resistance to prior therapy-Len+bortezomib refractory [Number; unit: participants]
  yes | 15 | 16 | 31
  no | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response, Analyzed Per International Myeloma Working Group Response Criteria
Description: All partial and complete responses must be confirmed with another efficacy assessment in no less than 4 weeks apart.
Time Frame: Efficacy assessments will be made after the first two cycles of therapy (approximately 56 days--each cycle is 28 days)
Measure: Number; unit: percentage of participants
Arm/Group | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle
Number analyzed (Participants) | 19 | 20
percentage of participants | 15.8 | 20.0

2. Primary Outcome: Percentage of Participants With Response, Analyzed Per International Myeloma Working Group Response Criteria
Description: All partial and complete responses must be confirmed with another efficacy assessment in no less than 4 weeks apart.
Time Frame: After the initial efficacy assessment at the completion of cycle 2 (at approximately 56 days), efficacy assessments will be made after every other cycle (approximately every 56 days).
Measure: Number; unit: percentage of participants
Arm/Group | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle
Number analyzed (Participants) | 19 | 20
percentage of participants
  cycle 4 | 15.8 | 40.0
  cycle 6 | 21.0 | 40.0
  cycle 8 | 21.0 | 45.0
  cycle 10 | 21.0 | 45.0
  cycle 12 | 21.0 | 45.0
  cycle 14 | 21.0 | 45.0

3. Secondary Outcome: To Compare the Effect of Continuous Versus Intermittent Regimens on F Actin Polymerization in Peripheral Blood Mononuclear Cells and Activation of Tumor Antigen-specific T Cells, as Well as Innate Lymphocytes (Natural Killer or Natural Killer T Cells).
Description: Correlation to be determined upon completion of study treatment
Time Frame: Research blood draw will be obtained at baseline, and at 2-4 hr (on day 1), 1 wk, and 4 wk after initiation of cycles 1 and 2.
Population: N/A: data were not collected on this outcome; initial F actin polymerization assay was unreliable and not reproducible; hence, this outcome could not be pursued.
Arm/Group | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Correlate Drug Induced Changes in F Actin Polymerization With Adverse Effects and Clinical Responses.
Description: Research bone marrow aspirate is obtained to assess response (optional, but recommended), and to document complete remission, if applicable. Correlation to be determined upon completion of study treatment
Time Frame: Research bone marrow aspirate is obtained at baseline and after completion of 2 cycles of therapy (approximately 56 days)
Population: The actin polymerization assay that was to be used for this outcome was not reproducible and data were not analyzed.
Arm/Group | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: To Correlate Drug Induced Changes in F Actin With Cytokine Profile.
Description: Correlation to be determined upon completion of study treatment
Time Frame: as for outcome 3
Population: The actin polymerization assay that was to be used for this outcome was not reproducible; hence, the cytokine profile of actin polymerized cells could not be pursued. Data were not analyzed.
Arm/Group | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle
Serious Adverse Events (participants affected / at risk) | 11/20 | 7/19
Other Adverse Events (participants affected / at risk) | 20/20 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle (N=20) | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle (N=19)
Febrile neutropenia (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 3 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Fever (General disorders) | 2 | 2
Syncope (Cardiac disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Cardiac disorders) | 1 | 0
Infection (Bacteremia) (Infections and infestations) | 1 | 0
Cardiac Disorders, other (Cardiac disorders) | 1 | 0
Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1
Hyperglycemia (Endocrine disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Infection (Other-Influenza) (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide 4 mg/d on 21 Days/28 Day Cycle (N=20) | Pomalidomide 2 mg/d on 28 Days/28 Day Cycle (N=19)
Anemia (Blood and lymphatic system disorders) | 10 | 6
Neutropenia (Blood and lymphatic system disorders) | 9 | 5
Leukopenia (Blood and lymphatic system disorders) | 15 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 6
Fatigue (General disorders) | 12 | 15
Nausea (General disorders) | 5 | 4
Vomiting (General disorders) | 2 | 2
AST increased (Hepatobiliary disorders) | 5 | 3
ALT increased (Hepatobiliary disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Dysguesia (Nervous system disorders) | 1 | 3
Edema Limbs (General disorders) | 3 | 2
Blurred vision (Nervous system disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Fever (General disorders) | 2 | 2
Anorexia (General disorders) | 5 | 2
Tremor (Nervous system disorders) | 4 | 3
Hyponatremia (Metabolism and nutrition disorders) | 6 | 3
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Pruritus (General disorders) | 5 | 3
Hot flashes (General disorders) | 5 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Dizziness (General disorders) | 4 | 2
Edema (General disorders) | 3 | 0
Creatinine increased (Renal and urinary disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Headache (Nervous system disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 3 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Soft tissue infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 2 | 1
Neuropathy (Nervous system disorders) | 3 | 1
Pain in extremity (General disorders) | 4 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Sore throat (General disorders) | 2 | 0
Bronchitis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Abdominal Pain (General disorders) | 1 | 1
Dry mouth (General disorders) | 1 | 1
Weight loss (General disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Hypertension (Cardiac disorders) | 1 | 1
Confusion (Nervous system disorders) | 1 | 1
Gait disturbance (Nervous system disorders) | 1 | 1
Productive cough (Infections and infestations) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Heightened sense of smell (Nervous system disorders) | 0 | 1
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Vertigo (Nervous system disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Insomnia (General disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 1
TSH increased (Endocrine disorders) | 0 | 1
T3 increased (Endocrine disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Periodontal disease (Infections and infestations) | 0 | 1
Flu-like symptoms (General disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Erectile dysfunction (General disorders) | 1 | 0
Libido decreased (Endocrine disorders) | 1 | 0
Muscle weakness, lower limb (Nervous system disorders) | 1 | 0
GERD (Gastrointestinal disorders) | 1 | 0
Presyncope (Cardiac disorders) | 1 | 0
Flatulence (General disorders) | 1 | 0
Nasal congestion (General disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Infection (other, oral) (Infections and infestations) | 1 | 0
Weight gain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes